CLINICAL TRIAL: NCT01537783
Title: A Randomized Trial to Evaluate a Staphylococcus Eradication Protocol for Patients Who Present to the Emergency Department With Cutaneous Abscess
Brief Title: Evaluation of a Staphylococcus Eradication Protocol for Patients Who Present to the ED With Cutaneous Abscess
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ED Staph Eradication
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Cutaneous Abscess
Keywords: abscess
MeSH Terms: conditions — Abscess | interventions — chlorhexidine gluconate; Mupirocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): In this arm, patients are treated with chlorhexidine scrubs once a day for 5 days and mupirocin nasal ointment inserted to both nostrils twice a day for 5 days. Both treatments are begun 7 days after enrollment, or when the abscess has healed fully if it has not healed by day 7.
  Interventions: Drug: Chlorhexidine gluconate; Drug: Mupirocin
- Standard of Care (No Intervention): In this arm, patients receive routine care of their abscess, which may or may not include either topical or oral antibiotics, at the discretion of the treating clinician.

INTERVENTIONS:
Drug: Chlorhexidine gluconate — Scrubs applied once a day for 5 days
  Other Names: Hibiclens
  Arms: Intervention group
Drug: Mupirocin — Nasal mupirocin applied topically to both nostrils twice a day for 5 days
  Other Names: Bactroban
  Arms: Intervention group

SUMMARY:
In this study, the investigators will enroll patients who present to the emergency department with abscesses to the study. The patients will be randomly selected to either have the standard of care, which includes the standard drainage of the abscess and then usually a follow-up visit to recheck the wound, or to have the standard of care plus instructions to use a topical scrub of a soap called chlorhexidine once a day for five days and twice daily application of a topical antibiotic ointment called mupirocin to the nasal passages for five days.

The investigators will then call back the patients at 7 days, 14 days (if in the treatment arm), 3 months and 6 months, to ask if they have had any recurrence of abscess formation. The study hypothesis is that the patients who have undergone the decontamination protocol will have fewer subsequent infections.

DETAILED DESCRIPTION:
Many people have heard of resistant "superbugs" which are causing worrisome infections in people around the world. One of these bacteria is called Methicillin Resistant Staphylococcus aureus (MRSA). Staph aureus is a pathogen that can lead to skin infections, but this newer strain is resistant to the standard antibiotic treatment that physicians used to render (usually penicillin-based). In addition, the community-acquired strain of MRSA is associated with creation of painful boils, or abscesses, which require patients to come and have a painful incision and drainage procedure in the ED. Soft tissue infections attributable to MRSA presenting to the ED and other ambulatory settings have increased at an alarming rate - from 32.1 to 48.1 visits per 1000 population when comparing data from the National Ambulatory Medical Care Survey and National Hospital Ambulatory Medical Care Survey from 1997 to 2005.

It is believed that MRSA is contracted from close contacts with other people who have the infection, and then it lives on the skin and nasal passages. For people who have recurrent skin infections, infectious disease experts sometimes recommend an "eradication" or "decolonization" protocol to try and kill off all of the MRSA. These protocols often involve a) a topical scrub to remove MRSA from the skin, b) a nasal antibiotic ointment to remove MRSA from the nasal passages, and occasionally c) an oral antibiotic. This procedure is usually recommended after seeing an infectious disease specialist, but to our knowledge, this has never been attempted from emergency department patients.

Therefore, in this study, the investigators will enroll patients who present to the emergency department with abscesses to the study. The patients will be randomly selected to either have the standard of care, which includes the standard drainage of the abscess and then usually a follow-up visit to recheck the wound, or to have the standard of care plus instructions to use a topical scrub of a soap called chlorhexidine once a day for five days and twice daily application of a topical antibiotic ointment called mupirocin to the nasal passages for five days.

The investigators will then call back the patients at 7 days, 14 days (if in the treatment arm), 3 months and 6 months, to ask if they have had any recurrence of abscess formation. The study hypothesis is that the patients who have undergone the decontamination protocol will have fewer subsequent infections.

Using a conservative estimate for the proportion of recurrence in the control group of 50%, a sample size of 50 (25 subjects in each group) will provide the investigators with 80% power to detect a statistically significant difference in the proportion of patients with recurrence between the treatment and control groups if the proportion of the treatment group with recurrent infection is 15%. If 60% of the control group experiences a recurrent infection, the study will have 80% power to detect a statistically significant difference if recurrence is observed in 23% of the treatment group.

If the hypothesis is true, it could greatly impact the care of patients who present with the ED with abscesses, and hopefully reduce the morbidity associated with having recurrent abscesses, including lost work and need to return for future painful incision and drainage procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years of age or older who present to our emergency department with a skin abscess which has undergone incision and drainage in which pus was present, and for whom the attending emergency physician is planning on discharging the patient home.

Exclusion Criteria:

* Abscesses resulting from insect or animal bites or intravenous drug use (both of which can be polymicrobial), chronic wounds (>2 weeks), wounds where no drainage was obtained in the course of the I&D, reported allergy to chlorhexidine or mupirocin, lack of ability to follow-up the patient (lack of phone number or stable address). Additionally, patients will be excluded who are of high acuity (unstable vital signs), in distress, with an insurmountable language barrier, intoxication (or other cause of altered mental status), presenting with acute psychiatric illness, are victims of possible sexual assault, or prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott G Weiner, MD, MPH, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Usual emergency department care
- Intervention: Usual emergency department care plus eradication protocol
Period: Overall Study
Arm/Group | Standard of Care | Intervention
Started | 25 | 25
Completed | 14 | 23
Not Completed | 11 | 2
Not completed — Lost to Follow-up | 11 | 2

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Standard emergency department care plus eradication protocol
- Standard of Care: Standard emergency department care
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Standard of Care | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: lost to followup
  years
    number analyzed (Participants) | 14 | 23 | 37
    (all) | 24.3 (5.2) | 35.4 (11.4) | 31.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: lost to followup
  Participants
    number analyzed (Participants) | 14 | 23 | 37
    Female | 9 | 12 | 21
    Male | 5 | 11 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of Cutaneous Abscess
Description: A patient's description that they have had another abscess since their index emergency department visit.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Standard of Care
Number analyzed (Participants) | 14 | 23
Participants | 5 | 7

ADVERSE EVENTS:
Arm/Group | Intervention Group | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
There were so many lost to follow-up patients in the intervention group that it is difficult to draw conclusions from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes